CLINICAL TRIAL: NCT02144246
Title: Contraceptive Hormones and Women With Cystic Fibrosis: Satisfaction and Effects on Disease
Brief Title: Contraceptive Hormones and Women With Cystic Fibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Courtney Schreiber, Family Planning Director, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 819889
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cystic Fibrosis Exacerbations While on and Off Hormonal Contraception
MeSH Terms: interventions — Moxifloxacin; Ethinyl Estradiol; norgestimate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-intervention (Other): Patients will act as their own controls. Will have no hormones for 3 months
  Interventions: Other: Non-hormonal period
- Post-intervention (Experimental): Ortho-cyclen (or a generic equivalent) which is Ethinyl estradiol/norgestimate, 0.035 mg/0.250 mg
  Interventions: Drug: Ortho-cyclen, Ethinyl estradiol/norgestimate, 0.035 mg/0.250 mg

INTERVENTIONS:
Other: Non-hormonal period
  Arms: Pre-intervention
Drug: Ortho-cyclen, Ethinyl estradiol/norgestimate, 0.035 mg/0.250 mg
  Other Names: Mononessa; Sprintec; Ethinyl estradiol/norgestimate, 0.035 mg/0.250 mg
  Arms: Post-intervention

SUMMARY:
Primary Objective Our primary objective in this study is to evaluate satisfaction of hormonal contraception in this sample of women and to evaluate the impact that this hormonal contraceptive has on cystic fibrosis (CF) disease in women with regular menstrual cycles accompanied by cyclic exacerbations.

We hypothesize:

1a) women with CF who perceive an overall benefit of hormonal contraception will be more satisfied than women with CF who do not perceive a benefit,

1b) women with CF who have cyclic exacerbations will have decreased Pseudomonas aeruginosa mucoidy conversion while using hormonal contraception,

1c) women with CF who have cyclic exacerbations will have improved patient-reported quality of life indices while on hormonal contraception, and

1d) women with CF who have cyclic exacerbations will have improvement in pulmonary function tests while on hormonal contraception.

Secondary Objective We plan to secondarily evaluate the cervical mucus of women with CF at the time of ovulation and compare it to that of healthy controls.

We hypothesize that women with CF have ovulatory cervical mucus similar to healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* female, reproductive age (18-40), cyclic CF exacerbations, regular menstrual cycles

Exclusion Criteria:

* pregnant, desires pregnancy, contra-indication to hormonal contraception, currently using hormonal contraception

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Satisfaction with contraception | 18 months
  Satisfaction overall
Exacerbation rate | 18 months
  Pseudomonas mucoidy conversion Quality of life Pulmonary function
Satisfaction with contraception | 18 months
  Satisfaction overall measured by a visual analog scale 0-10

SECONDARY OUTCOMES:
Cervical Mucus | 3 months
  Cervical mucus of CF patients relative to healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States